CLINICAL TRIAL: NCT04926883
Title: Clinical Performance of Sonic-Activated High Viscosity Bulk-Fill Resin Composite in Comparison to Conventional Bulk-Fill Resin Composite Restorations in Posterior Teeth: A Randomized Controlled Clinical Study.
Brief Title: Comparison Between Sonic Fill and X-tra Fill in Clinical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ashraf Aref, PhD candidate, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Bulkfill2021
Record Dates: First submitted 2021-06-03; First posted 2021-06-15 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: SonicFill Clinical Performance; Sonicated Bulk-fill Resin Composite
Keywords: bulk-fill; resin composite; sonicfill; clinical performance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonic fill (Active Comparator)
  Interventions: Other: bulk-fill composite resin restorations
- X-tra fill (Active Comparator)
  Interventions: Other: bulk-fill composite resin restorations

INTERVENTIONS:
Other: bulk-fill composite resin restorations — bulk-fill composite resin restorations up to 5mm layer thickness

SUMMARY:
The present study aims to evaluate a 2-years clinical performance of sonic-activated bulk-fill resin composite material (sonic fill) in comparison to conventional bulk-fill resin composite (X-tra fill) as posterior restorations. The null hypothesis is that sonic-activated bulk-fill resin composite restoration shows no difference when compared to conventional bulk-fill resin composite in clinical performance over 2-years evaluations based on clinical assessment.

DETAILED DESCRIPTION:
Restorations will be evaluated 1 week after placement (Baseline - T0), 3 months (T1), 6 months (T2), 1-year (T3) and 2-years (T4) of clinical service by blinded calibrated examiner using modified United States Public Health Service (USPHS) criteria where score A (Alpha) stands for the clinically ideal restoration. Score B (Bravo) is a clinically acceptable situation except for secondary caries. Score C (Charlie) indicates clinically unacceptable restorations that must be replaced.

The restorations will also be evaluated using revised FDI criteria with five grades for each criterion; scores 1 to 3 indicated clinically acceptable restorations, and scores 4 and 5 summarized clinically unacceptable situations indicating repair (score 4) or replacement (score 5).

ELIGIBILITY:
Inclusion Criteria:

* They should have an acceptable oral hygiene level.

  * Presence of at least two posterior carious lesions to be restored with two different types of composite.
  * The two materials should be used in approximately the same sized lesions or within the same extension.
  * Age range between 18 and 45 years.
  * A good likelihood of recall availability.

Exclusion Criteria:

* Severe or active periodontal or carious disease.
* Heavy bruxism or a traumatic occlusion.
* Patients with a compromised medical history or had received therapeutic irradiation to the head and neck region.
* Alcoholic and smoker patients.
* Patients had participated in a clinical trial within 6 months before commencement of this trial.
* Patients unable to return for recall appointment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
change in clinical performance | 1 week, 3 months, 6 months, 12 months
  restorations' evaluation for retention, color matching, marginal discoloration, marginal adaptation, secondary caries, surface texture, anatomic form.
  Score A (Alpha) stands for the clinically ideal restoration. Score B (Bravo) is a clinically acceptable situation except for secondary caries. Score C (Charlie) indicates clinically unacceptable restorations that must be replaced. Also will be scored from 1 to 5 , which 1 to 3 indicated clinically acceptable restorations, and scores 4 and 5 summarized clinically unacceptable situations indicating repair (score 4) or replacement (score 5).

SECONDARY OUTCOMES:
change in post-operative pain using modified Visual Analogue Scale (VAS) | daily for 1 week
  The patients will be asked to record their pain level on modified Visual Analogue Scale (VAS) from 0 to 10, where 10 means sever pain, for 1 week.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

REFERENCES:
- [Derived] Aref A, Abd-Elhakim S, Riad M. 24-month randomized controlled clinical trial assessment of surface texture, color stability, and marginal discoloration of sonic activated bulk-fill resin composite according to USPHS and FDI criteria. BMC Oral Health. 2025 Jul 26;25(1):1261. doi: 10.1186/s12903-025-06611-0. PMID 40713556